CLINICAL TRIAL: NCT05467449
Title: DxFLEX ClearLLab 10C US-IVD Clinical Study Protocol - Clinical Laboratory
Brief Title: DxFLEX 10C Clinical Study
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C76895
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Hematologically normal: Based on immunophenotyping
  Interventions: Device: DxFLEX 10C
- Hematologically abnormal: Based on immunophenotyping
  Interventions: Device: DxFLEX 10C

INTERVENTIONS:
Device: DxFLEX 10C — A device combining flow cytometry and reagents for immunophenotyping analysis

SUMMARY:
A multi-center method comparison study is designed per CLSI-EP09 A3. This study compares the qualitative immunophenotype agreement between DxFLEX and Navios EX to demonstrate the accuracy of the DxFLEX-10C system. A series of precision studies will be conducted with each focusing on different aspects of the DxFLEX-10C system.

ELIGIBILITY:
Inclusion Criteria: Patient specimens targeted for this study will be residual samples with sufficient volume from whole blood, bone marrow, and lymph node meeting the following criteria:

1. Specimens from new cases or follow up patients for myeloid/lymphoid FCI testing.
2. Hematologically abnormal specimens
3. Subjects of any range, ethnicities, and racial backgrounds
4. Specimens from patients with the following medical indications presenting for testing by flow cytometry based on the Bethesda Consensus Guidelines.

Exclusion Criteria:

There are two (2) groups of exclusion criteria to detail the specimens that should not be counted for the study:

1. Pre-analytical/Pre-screen exclusion criteria
2. Post-acquisition exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intended L&L population
Sampling Method: Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Flow immunophenotyped normal and abnormal | immediately after the analysis
  Based on WHO guidelines for Leukemia & Lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Guoyan Cheng, PhD, Study Director — Beckman Coulter, Inc.
Locations (6):
- United States (4):
  - NeoGenomics Laboratories, Aliso Viejo, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Quest Diagnostics, Lewisville, Texas
  - PhenoPath Laboratories, PLLC, Seattle, Washington
- London Health Sciences Centre, London, Ontario, Canada
- Munich Leukemia Laboratory (MLL), Munich, Germany

IPD SHARING:
Plan to Share IPD: No